CLINICAL TRIAL: NCT00945516
Title: Newly Designed Fully Covered Metal Stent for the Benign Biliary Stricture: Prospective Randomized Study
Brief Title: Newly Designed Fully Covered Metal Stent for the Benign Biliary Stricture
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Jung Sin Lee / the director of a center, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2009-0233
Record Dates: First submitted 2009-07-20; First posted 2009-07-24 (Estimated); Last update posted 2010-10-19 (Estimated); Status verified 2010-10

CONDITIONS: Bile Duct Disease
Keywords: Metal stent; Bile duct stricture; Stent migration; Feasibility; Safety; Removability
MeSH Terms: conditions — Bile Duct Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Flared end FCSEMS (Active Comparator): Flared end FCSEMS will be inserted for the benign bile duct stricture.
  Interventions: Device: Bona stent® (Flared end FCSEMS)
- Anchoring FCSEMS (Active Comparator): Anchoring FCSEMS will be inserted for benign bile duct stricture
  Interventions: Device: Hanarostent® (Anchoring FCSEMS)

INTERVENTIONS:
Device: Bona stent® (Flared end FCSEMS) — Flared end FCSEMS for benign bile duct stricture will be inserted with ERCP.
  Other Names: Bona stent® (Sewoon medical Co., LTD., Seoul, Korea)
  Arms: Flared end FCSEMS
Device: Hanarostent® (Anchoring FCSEMS) — Anchoring FCSEMS for benign bile duct stricture will be inserted with ERCP.
  Other Names: Hanarostent® (M.I.Tech, Seoul, Korea)
  Arms: Anchoring FCSEMS

SUMMARY:
The purpose of this study is to determine the feasibility, easy removability, safety, and migration rate of flared end fully covered self-expanding metal stent (FCSEMS) and anchoring FCSEMS for benign biliary stricture.

DETAILED DESCRIPTION:
Benign biliary strictures (BBS) are usually managed with plastic stents, whereas placement of uncovered metallic stents has been associated with failure related to mucosal hyperplasia. Fully covered self-expanding metal stent(FCSEMS) placement was reported as a useful method for BBS. However, stent migration was a frequent complication of CSEMS placement. Recently, flared end FCSEMS was developed to decrease stent migration, and anchoring CSEMS was newly developed.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years old
* Patient with benign bile duct stricture

Exclusion Criteria:

* No written informed consent
* Malignant biliary obstruction
* Patients with uncorrectable severe coagulopathy
* Patients with severe cardiopulmonary disease precluding sedation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2009-01; Primary Completion 2010-04 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Stent migration rate | one year

SECONDARY OUTCOMES:
Feasibility (Technical success rate and functional success rate) | one year
Safety (Procedure related early complications occurred within one month and late complications occurred one month after the procedure) | one year
Removability | one year

CONTACTS AND LOCATIONS:
Overall Officials: Do Hyun Park, MD, PhD, Study Director — Department of Gastroenterology, University of Ulsan College of Medicine, Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, Seoul, South Korea

REFERENCES:
- [Derived] Park DH, Lee SS, Lee TH, Ryu CH, Kim HJ, Seo DW, Park SH, Lee SK, Kim MH, Kim SJ. Anchoring flap versus flared end, fully covered self-expandable metal stents to prevent migration in patients with benign biliary strictures: a multicenter, prospective, comparative pilot study (with videos). Gastrointest Endosc. 2011 Jan;73(1):64-70. doi: 10.1016/j.gie.2010.09.039. PMID 21184871